CLINICAL TRIAL: NCT03470116
Title: MILAR, is a Controlled, Randomised, Comparative, Prospective, Multi-center, Superiority French Clinical Trial Comparing the MacGrath MAC Videolaryngoscope and the MacIntosh Laryngoscope for Oro-tracheal Intubation by Patients With Less Than 2 Criteria of Difficult Intubation in Elective Surgery.
Brief Title: Comparison Between the MacGrath MAC Videolaryngoscope and the MacIntosh Laryngoscope for Oro-tracheal Intubation for Patients With Less Than 2 Criteria of Difficult Intubation in Elective Surgery.
Acronym: MILAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHRO-2017-13
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Laryngoscopy
Keywords: MacGrath MAC; curarization; intubation; MacIntosh; laryngoscope
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MacGrath MAC video laryngoscopy (Experimental): Patients will benefit MacGrath MAC video laryngoscopy for intubation after curarization
  Interventions: Device: Laryngoscopy with Mac Grath
- direct laryngoscopy (Active Comparator): Patients will benefit direct laryngoscopy for intubation after curarization
  Interventions: Device: direct laryngoscopy

INTERVENTIONS:
Device: Laryngoscopy with Mac Grath — Patients of this group will benefit MacGrath MAC video laryngoscopy for intubation after curarization
  Arms: MacGrath MAC video laryngoscopy
Device: direct laryngoscopy — Patients of this group will benefit direct laryngoscopy for intubation after curarization
  Arms: direct laryngoscopy

SUMMARY:
The MILAR trial is a multicenter randomised , prospective, controlled, single-blind, superiority French clinical trial, with a 1: 1 distribution of patients to compare intubation during the first laryngoscopy between the MacGrath MAC videolaryngoscope and the MacIntosh laryngoscope for patients with less than 2 criteria of difficult intubation in elective surgery.

DETAILED DESCRIPTION:
Tracheal intubation is a common procedure in the operating room to secure the airway in patients receiving muscle relaxants .

Two devices are currently used for this purpose with various indications: the French Society of Anesthesia and Resuscitation (SFAR) recommends a direct laryngoscopy with MacIntosh blade in first intention for patients with less than 2 criteria of difficult intubation (ID). The SFAR recommends first-line video laryngoscopy in patients with two or more criteria of difficult intubation. Video laryngoscopy improves glottic vision, difficult intubation score, and intubation success rate at the first attempt, compared to the direct laryngoscopy with a Macintosh blade.

Currently, it is estimated that 15% of direct laryngoscopies with a MacIntosh blade result in failure of orotracheal intubation (IOT) on first attempt, whereas tracheal intubation with a video laryngoscopy is a better solution to secure the airway.

Our hypothesis in this study is that the MacGrath MAC videolaryngoscope allows to intubate at the first laryngoscopy 91% of patients with less than 2 difficult intubation criteria, against the expected 85% with the MacIntosh blade.

ELIGIBILITY:
Inclusion Criteria:

less than 2 criteria of difficult intubation admitted to the operating theater for scheduled surgery requiring orotracheal intubation after curarization - informed consent

Exclusion Criteria:

* pregnancy
* age < 18
* contraindication to oro-tracheal intubation
* emergency surgery
* thoracic surgery
* naso-tracheal intubation
* patient protected by law
* patient not affiliated to french social security
* BMI> 45kg / m²
* Predicted patient with difficult intubation

Patients considered to be predisposed to difficult intubation are those with a history of difficult intubation, or with 2 criteria among:

* Mallampati 3 or 4
* Thyroid-chin distance <65mm
* Mouth opening <35mm
* Spinal extension less than 90 °
* Retrognathism with Negative Lip Test
* Morbid obesity with BMI> 35kg / m²
* Obstructive Sleep Apnea Syndrome with choker> 45cm
* Diabetic with sign of the positive prior
* Head and Neck Pathology

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Successful first attempt intubation after curarization | 2 minutes
  The primary endpoint is the success of tracheal intubation by anesthesiologists or registrated nurse anesthetists on exposure to first laryngoscopy, confirmed by three identical capnographic curves on the monitor.

SECONDARY OUTCOMES:
Presence of glottal exposure during the first laryngoscopy | 2 minutes
  presence or absence of glottal exposure during the first laryngoscopy
Use of a second laryngoscopy | 2 minutes
  Use or not of a second laryngoscopy
Type of laryngoscope used in second laryngoscopy | 2 minutes
  If second laryngoscopy is practice, name of second laryngoscope
Use of a mandrel | 2 minutes
  use or not of a mandrel
Use of a supra-glottal device | 2 minutes
  Use or not of a supra-glottal device
Use of a fibreoptic | 2 minutes
  Use or not of a fibreoptic
Use of a transtracheal oxygenation device | 2 minutes
  Use or not of a transtracheal oxygenation device
Presence of desaturations <92% during laryngoscopy | 2 minutes
  presence or absence of desaturation
number of esophageal intubation | 2 minutes
Pharyngeal lesions / bleeding | 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: MFAM Willy Serge, MD, Principal Investigator — ORLEANS REGIONAL HOSPITAL CENTER; SINDA Patrick, MD, Principal Investigator — CHARTRES HOSPITAL CENTER
Locations (2):
- France (2):
  - Chartres Hospital Center, Chartres
  - Orleans Hospital Center, Orléans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook TM, Woodall N, Harper J, Benger J; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 2: intensive care and emergency departments. Br J Anaesth. 2011 May;106(5):632-42. doi: 10.1093/bja/aer059. Epub 2011 Mar 29. PMID 21447489
- [Background] Hasegawa K, Shigemitsu K, Hagiwara Y, Chiba T, Watase H, Brown CA 3rd, Brown DF; Japanese Emergency Medicine Research Alliance Investigators. Association between repeated intubation attempts and adverse events in emergency departments: an analysis of a multicenter prospective observational study. Ann Emerg Med. 2012 Dec;60(6):749-754.e2. doi: 10.1016/j.annemergmed.2012.04.005. Epub 2012 Apr 28. PMID 22542734
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Sakles JC, Javedani PP, Chase E, Garst-Orozco J, Guillen-Rodriguez JM, Stolz U. The use of a video laryngoscope by emergency medicine residents is associated with a reduction in esophageal intubations in the emergency department. Acad Emerg Med. 2015 Jun;22(6):700-7. doi: 10.1111/acem.12674. Epub 2015 May 20. PMID 25996773
- [Background] Kaplan A, Goksu E, Yildiz G, Kilic T. Comparison of the C-MAC Videolaryngoscope and Rigid Fiberscope with Direct Laryngoscopy in Easy and Difficult Airway Scenarios: A Manikin Study. J Emerg Med. 2016 Mar;50(3):e107-14. doi: 10.1016/j.jemermed.2015.06.070. Epub 2015 Dec 22. PMID 26725922
- [Background] Ruetzler K, Imach S, Weiss M, Haas T, Schmidt AR. [Comparison of five video laryngoscopes and conventional direct laryngoscopy : Investigations on simple and simulated difficult airways on the intubation trainer]. Anaesthesist. 2015 Jul;64(7):513-9. doi: 10.1007/s00101-015-0051-5. Epub 2015 Jul 15. German. PMID 26174747